CLINICAL TRIAL: NCT01760551
Title: Correlation Between the American Medical Association Guides to the Evaluation of Permanent Impairment and the Medical Outcomes Study 36-Item Short Form.
Status: Completed | Type: Observational
Sponsor: JointResearch (Other)
Collaborators: McMaster University (Other); Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Sponsor
Other Study IDs: JR201201
Record Dates: First submitted 2012-12-28; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Trauma
Keywords: Fracture; Trauma; impairment
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients assessed with AMA guide fifth edition
- Patients assessed with AMA guide sixth edition

SUMMARY:
The American Medical Association's (AMA) Guides to the Evaluation of Permanent Impairment is used to rate loss of function and determine compensation and ability to work after injury or illness. The AMA Guides are used by many different systems to determine compensable levels of impairment. However, there are few studies that evaluate reliability or construct validity. (1) In the professional community there exists considerable controversy regarding the accuracy and usefulness of the AMA Guides. (2,3) Commentaries have noted that the AMA Guides do not provide a valid, reliable, evidence-based system for the rating of impairments. (4) Some have argued that the impairment ratings do not reflect an individual's actual loss of function and quality of life (QOL). The AMA guides 5th edition was based on loss of range of motion (ROM). The new 6th edition of the AMA guides is based on diagnosis and inclusion of functional outcomes assessments in the determination of impairment ratings. (5) In the orthopaedic literature the use of patient-derived, objective outcome measures has substantially expanded QOL instruments are categorized as general health or as condition-specific questionnaires. The Medical Outcomes Study 36-Item Short Form (SF-36) is a general health-based survey of quality of life. It has been validated and is used widely across medical disciplines. (6) The SF-36 was constructed to survey health status in the Medical Outcomes Study. It was designed for use in clinical practice and research, health policy evaluations, and general population surveys. The SF-36 was constructed for self-administration by persons 14 years of age and older, and for administration by a trained interviewer in person or by telephone. (7) The SF-36 is perhaps the most widely used health-related quality of life (HRQoL) survey instrument in the world today. It is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. (8) The aim of this study is to determine the amount of correlation between the by orthopaedic surgeon objectively calculated percentage of impairment scored by the American Medical Association guides to the evaluation of permanent impairment and the by patient subjectively indicated health-related quality of life scored by the SF-36.

Hypotheses: Because of and inclusion of functional outcomes assessments in the determination of impairment ratings the AMA guide 6th edition will have a better correlation with the SF-36. The 6th edition of the AMA guide is based on diagnosis en yield lower impairment percentages than the AMA guide 5th edition that is based on loss of ROM. The SF-36 will have better correlation with the impairment ratings for lower extremities injuries than for upper extremities because it is less valid for the upper extremities.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who have had a medical legal examination

Exclusion Criteria:

* exclusion if there is no calculation of the percentage of impairment by the American Medical Association guides to the evaluation of permanent impairment.

Age under 14 years

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have had a medical legal examination by an orthopaedic surgeon working at "Orthopedisch Expertise Centrum" and have completed a to Dutch translated SF-36 form.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fifth or Sixth AMA Guide impairment rating | Once at assessment of impairment consultation 1hour
  https://catalog.ama-assn.org/Catalog/product/product_detail.jsp?productId=OP025400
  https://catalog.ama-assn.org/Catalog/product/product_detail.jsp?productId=prod920005

SECONDARY OUTCOMES:
RAND 36 | Once at assessment during impairment consultation for app 1hour
  http://www.ncbi.nlm.nih.gov/pubmed/19364637

OTHER OUTCOMES:
DASH | Once at assessment during impairment consultation for app 1hour
  http://www.ncbi.nlm.nih.gov/pubmed/18473398

CONTACTS AND LOCATIONS:
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands